CLINICAL TRIAL: NCT05587296
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Study to Investigate Efficacy and Safety of Elinzanetant for the Treatment of Vasomotor Symptoms Induced by Adjuvant Endocrine Therapy, Over 52 Weeks and Optionally for an Additional up to 2.5 Years in Women With Hormone-receptor Positive Breast Cancer:
Brief Title: A Study to Learn More About How Well Elinzanetant Works and How Safe it is Compared to Placebo for the Treatment of Hot Flashes Caused by Anti-cancer Therapy in Women With, or at High Risk for Developing Hormone-receptor Positive Breast Cancer
Acronym: OASIS-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21656; 2023-508265-33-00 (Registry Identifier: CTIS (EU)); 2022-000095-18 (EudraCT Number)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms Caused by Adjuvant Endocrine Therapy in Women With, or at High Risk for Developing Hormone-receptor Positive Breast Cancer; Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Elinzanetant (BAY3427080) (Experimental): Participants will receive 120 mg elinzanetant orally once daily.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Placebo (Placebo Comparator): Participants will receive matching placebo orally once daily for 12 weeks, followed by 120 mg elinzanetant orally once daily
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — 120 mg elinzanetant orally once daily
Drug: Placebo — Matching placebo orally once daily
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to treat women with, or at high risk for developing hormone-receptor positive breast cancer, who have vasomotor symptoms (VMS), a condition of having hot flashes caused by anti-cancer therapy.

VMS, also called hot flashes, are very common medical problems in women with hormone-receptor (HR)-positive breast cancer, who are receiving anti-cancer therapy. HR-positive breast cancer is a type of breast cancer, which has hormone-receptors (proteins) for female sex hormones estrogen and/or progesterone. These hormone-receptors may attach to hormones like estrogen and progesterone and thereby help cancer cells to grow and to spread. Treatments that stop these hormones from attaching to these receptors are currently used to slow or stop the growth of HR-positive breast cancer.

It is already known that women with HR-positive breast cancer benefit from this treatment. However, hot flashes are common medical problems related to this therapy. They negatively affect quality of life of many women and may lead to discontinuation (stopping) of this therapy.

The study treatment, elinzanetant is being developed to treat hot flushes. It works by blocking a substance called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes.

The main purpose of this study is to learn more about how well elinzanetant helps to treat hot flashes caused by anti-cancer therapy in women with or at high risk for developing HR-positive breast cancer compared to placebo. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

To answer this, the doctors will ask the participants to record information about their hot flashes before treatment start and at certain time points during the treatment in an electronic diary. The researchers will then assess possible average changes in number and severity of hot flashes after 4 and 12 weeks of treatment.

To see how safe elinzanetant is compared to placebo. The study will collect information about the number of participants who have medical problems after taking treatment.

The study participants will be randomly (by chance) assigned to 2 treatment groups, A and B. The participants from treatment group A will take elinzanetant. The participants from treatment group B will start with placebo and then switch to elinzanetant.

All participants will continue taking the anti-cancer therapy they have been using when entering the study.

Dependent on the treatment group, the participants will either take elinzanetant or placebo as capsules by mouth once a day. After 12 weeks, the participants who have initially received placebo will switch to take elinzanetant for the remaining 40 weeks.

Each participant will be in the study for approximately 62 weeks. The treatment duration in the study will be 52 weeks. There will be up to 12 visits to the study site and 6 phone calls in between. Participants who completed the 52 weeks treatment phase, will be offered to continue treatment for another up to 2.5 years. Visit frequency: every 24 weeks until week 152.

During the study, the participants will:

* record information about their hot flashes
* answer questions about their quality of life and other symptoms.

The doctors and their study team will:

* check the participants health and vital signs
* take blood and urine samples
* examine heart health using electrocardiogram (ECG)
* examine pelvic organs like womb or ovaries using a trans vaginal ultrasound scan to see images of these organs
* make images of the breast using x-ray (mammogram), a type of radiation that passes through the body to make images of the inside and/or by using ultrasound (if applicable)
* check the health of the participant's cervix (neck of the womb) by taking a small sample of cells (smear test) for an analysis called cervical cytology (if applicable)
* take an endometrial biopsy, a small piece of tissue from the lining of the womb (called the endometrium) for analysis.
* ask the participants questions about what medicines they are taking and if they are having adverse events.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

About 4 weeks after the participants take their last treatment, the study doctors and their team will check the participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 70 years of age inclusive, at the time of signing the informed consent.
* Women experiencing vasomotor symptoms (VMS) caused by adjuvant endocrine therapy that they are expected to use for the duration of the study

  * Tamoxifen with or without the use of gonadotropin-releasing hormone (GnRH) analogues or
  * Aromatase inhibitors with or without the use of GnRH analogues
* Women must have

  * a personal history of hormone-receptor positive breast cancer or
  * a high risk for developing breast cancer.
* Participant has completed Hot Flash Daily Diary (HFDD) for at least 11 days during the two weeks preceding baseline visit, and participant has recorded at least 35 moderate to severe hot flash (HF) (including night-time HF) over the last 7 days that the HFDD was completed (assessed at the Baseline Visit).
* Contraceptive use by [women except for post-menopausal women or Women of Non childbearing potential (WONCBP)] should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Initial diagnosis of metastatic hormone-receptor positive breast cancer (stage IV) or recurrence under adjuvant endocrine therapy of hormone-receptor positive breast cancer.
* Current or history (except complete remission for 5 years or more prior to signing informed consent) of any malignancy, except for hormone-receptor positive breast cancer (Stage 0-III), basal and squamous cell skin tumors.
* Surgery or non-surgical (e.g., chemotherapy, radiotherapy, immunotherapy) treatment for breast cancer within the last 3 months prior to signing informed consent (except use of tamoxifen, aromatase inhibitors, GnRH analogues).
* Any clinically significant prior or ongoing history of arrhythmias, heart block and QT prolongation either determined through clinical history or on electrocardiogram (ECG) evaluation.
* Any active ongoing condition that could cause difficulty in interpreting VMS such as: infection that could cause pyrexia, pheochromocytoma, carcinoid syndrome.
* Any unexplained vaginal bleeding.
* Mammogram with clinically relevant malignant or suspicious findings that will require surgery, radiotherapy or chemotherapy as per local guidelines (mammogram should not be older than 12 months prior to signing informed consent). If a mammogram is not possible after partial mastectomy an ultrasound could be performed instead.
* Disordered proliferative endometrium, endometrial hyperplasia, polyp, or endometrial cancer diagnosed based on endometrial biopsy during screening.
* Current arterial or venous vascular event (e.g., Myocardial infarction (MI), Transient ischemic attack (TIA), stroke, deep vein thrombosis (DVT), i.e., within the last 6 months prior to signing informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2028-06-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (102):
- Austria (3):
  - Medical University of Graz | Division of Gynecology and Obstetrics, Graz, Styria
  - MedUni Innsbruck | Brust Gesundheit Zentrum, Innsbruck, Tyrol
  - AKH Wien | Allg. Gynaekologie & gynaekologische Onkologie, Vienna
- Belgium (8):
  - ZAS Augustinus - Gynaecology department, Wilrijk, Antwerpen
  - Hôpital Erasme/Erasmus Ziekenhuis, Brussels
  - CHU Saint-Pierre/UMC Sint-Pieter, Bruxelles - Brussel
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - Ziekenhuis Oost-Limburg - Gynecology Department, Genk
  - Ghent University Hospital | Women's Clinic Department, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Femicare vzw | Tienen, BE, Tienen
- Canada (2):
  - The Ottawa Hospital - Riverside Campus, Ottawa, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal (CRCHUM), Montreal, Quebec
- Finland (5):
  - Docrates Mehiläinen Syöpäsairaala, Helsinki
  - Mehiläinen Kuopio, Kuopio
  - Lääkärikeskus Gyneko Oy, Oulu
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS), Tampere
  - Vaasa Central Hospital, Vaasan keskussairaala - Syöpätaudit, Vaasa
- France (9):
  - ICO Site Paul Papin - Angers - Service Oncologie, Angers
  - Institut Bergonie - Unicancer Nouvelle Aquitaine, Bordeaux
  - Centre de Lutte Contre le Cancer François Baclesse - Service Pathologie mammaire, Caen
  - UNICANCER - Centre Leon-Berard (CLB) - Medical oncology, Lyon
  - Institut du Cancer de Montpellier - Val d'Aurelle - Service Oncogynecologie et senologie, Montpellier
  - Hôpital Saint Louis, Paris
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Tenon - Gynecologie Obstetrique Medecine de la Reproduction, Paris
  - Institut de Cancerologie Ouest - Saint-Herblain - Service gynecologie medicale, Saint-Herblain
  - ICANS - Institut de Cancerologie de Strasbourg Europe, Strasbourg
- Germany (12):
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Eberhard-Karls-Universität Tübingen, Tübingen, Baden-Wurttemberg
  - Synexus Frankfurt Clinical Research Centre, Frankfurt am Main, Hesse
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Praxis Hr. Dr. S. Fiedler, Aachen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bergisch Gladbach - Gynäkologi, Bergisch Gladbach, North Rhine-Westphalia
  - Gynäkologisches Zentrum Bonn, Bonn, North Rhine-Westphalia
  - Frauenärzte am Schloss Borbeck, Essen, North Rhine-Westphalia
  - Medplus Nordrhein, Krefeld, North Rhine-Westphalia
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - Frauenarztpraxis Dr. Inka Kiesche, Halle, Saxony-Anhalt
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Axon Kft., Kecskemét
  - Szabolcs Szatmr Bereg County University Teaching Hospital | Andras Jasa Teaching Hospital - Oncology, Nyíregyháza
  - Rub-Int Noi Egeszsegcentrum, Székesfehérvár
- Ireland (6):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - St James' Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - University College Hospital Galway, Galway
  - University Hospital Waterford, Waterford
- Israel (6):
  - Assuta Ashdod Public Hospital (R.A), Ashdod
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Health Corporation of Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Azienda Ospedaliera Universitaria Federico II Di Napoli - DAI Materno Infantile, Napoli, Campania
  - Azienda Ospedaliero Universitaria di Modena_Policlinico - Oncologia, Modena, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Ginecologia Oncologica, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino - Clinica ostetrica e ginecologica, Genoa, Liguria
  - Istituto Europeo di Oncologia s.r.l - Ginecologia Preventiva, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo - Ostetricia e Ginecologia, Pavia, Lombardy
  - Azienda Ospedaliera Ordine Mauriziano Di Torino - Ostetricia e Ginecologia, Turin, Piedmont
  - Careggi University Hospital - Ostetricia e Ginecologia, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Verona_Borgo Trento - Ostetricia e Ginecologia B, Verona, Veneto
- Kazakhstan (2):
  - Kazakh Institute of Oncology and Radiology - Department of Gynecology, Almaty
  - Multidisciplinary Medical Center of the Akimat of Astana - Department of Chemotherapy No1, Astana
- Poland (8):
  - Gabinet Ginekologiczny Janusz Tomaszewski, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - NZOZ MEDEM Wilk Sp. j., Katowice
  - Pratia McM Kraków, Krakow
  - Prywatny Gabinet Lekarski Ginekologia, Poloznictwo i Ultr., Lodz
  - Salve Medica Sp. z o.o. SP.K., Lodz
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
- Portugal (10):
  - Luz Saude | Hospital Beatriz Angelo - Centro de Investigacao Clinica, Loures, Lisbon District
  - Centro Clinico Academico Braga | Braga, Portugal, Braga
  - Centro Hospitalar e Universitario de Coimbra, E.P.E. | Department of Gynecology, Coimbra
  - Fundacao Champalimaud | Centro Clinico Champalimaud - Unidade Investigacao Clinica, Lisbon
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
  - CHULN - H. Sta.Maria (Centro de Investigacao Clinica), Lisbon
  - Centro Hospitalar Universitario do Porto, Porto
  - Companhia Uniao Fabril | Hospital CUF Porto - Clinical Trials Department, Porto
  - CHUSJ - Hospital Sao Joao, Porto
- Romania (5):
  - Sc Oncolab Srl, Craiova, Dolj
  - S.C. Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov
  - S.C. Quantum Medical Center SRL, Bucharest
  - Spitalul Clinic Filantropia, Bucharest
  - S.C Ovidius Clinical Hospital SRL - Oncology Department, Ovidiu
- Spain (8):
  - Complexo Hospitalario Universitario De Santiago | Oncologia, Santiago de Compostela, A Coruña
  - La Zarzuela University Hospital | Ginecologia, Aravaca, Madrid
  - Hospital del Mar I Ginecologia, Barcelona
  - Hospital Universitario Virgen De Las Nieves | Oncologia Medica, Granada
  - Hospital General Universitario Gregorio Maranon | Oncologia, Madrid
  - Hospital Universitario Virgen Del Rocio S.L. | Oncologia, Seville
  - Hospital Clinico Universitario De Valencia | Ginecologia, Valencia
  - Hospital General Universitario De Valencia | Ginecologia, Valencia
- United Kingdom (5):
  - Imperial College Healthcare NHS Trust| Queen Charlotte's and Chelsea Hospital - Gynaecology, London, Greater London
  - Liverpool Women's NHS Foundation Trust | Liverpool Women's Hospital - Gynaecology, Liverpool, Merseyside
  - NHS Greater Glasgow and Clyde | Glasgow Royal Infirmary - Gynaecology, Glasgow, Scotland
  - Surrey and Sussex Healthcare NHS Trust - East Surrey Hospital - Gynaecology, Redhill, Surrey
  - NHS Grampian | Aberdeen Royal Infirmary - Gynaecology, Aberdeen

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Cardoso F, Parke S, Brennan DJ, Briggs P, Donders G, Panay N, Haseli-Mashhadi N, Block M, Caetano C, Francuski M, Haberland C, Laapas K, Seitz C, Zuurman L. Elinzanetant for Vasomotor Symptoms from Endocrine Therapy for Breast Cancer. N Engl J Med. 2025 Aug 21;393(8):753-763. doi: 10.1056/NEJMoa2415566. Epub 2025 Jun 2. PMID 40454634
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 97 study centers, predominantly in Europe and at several centers in Canada, Israel, Kazakhstan and United Kingdom starting 14-Oct-2022 (first participant first visit), reaching primary completion on 29-Jan-2024.
Pre-assignment Details: Out of 758 screened participants, 474 were randomized.
Groups:
- Elinzanetant (BAY3427080): Participants received 120 mg elinzanetant orally once daily for 52 weeks
- Placebo - Elinzanetant (BAY3427080): Participants received placebo orally once daily for the first 12 weeks. 120 mg elinzanetant was administered from Week 13 to 52.
Period: Overall Study
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Started | 316 | 158
Completed | 262 | 133
Not Completed | 54 | 25
Not completed — Adverse Event | 15 | 7
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 14 | 4
Not completed — miscellaneous | 3 | 6
Not completed — Did not complete study treatment but completed post-treatment phase/follow-up | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080) | Total
Number analyzed (Participants) | 316 | 158 | 474
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (7.5) | 51.5 (6.7) | 51.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 158 | 474
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 289 | 143 | 432
  Unknown or Not Reported | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe Hot Flashes (HF) From Baseline to Week 4 (Assessed by Hot Flash Daily Diary [HFDD])
Description: Participants' assessments of HF were recorded electronically twice daily using the sponsor developed Hot Flash Daily Diary (HFDD). The HFDD was completed in the morning after waking up (morning diary) and each evening at bedtime (evening diary) on the hand-held device. The HFDD items assessed the number of mild, moderate, and severe HF experienced during the day and during the night. Mild HF was defined as a "sensation of heat without sweating", moderate HF was defined as a "sensation of heat with sweating, but able to continue activity", and severe HF was defined as a "sensation of heat with sweating, causing cessation (stopping) of activity". Mean daily frequency is calculated as total number of moderate to severe HF during that week divided by the total number of available days with data during that week.
Time Frame: Baseline to Week 4
Population: FAS
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
hot flashes per day
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 11.41 (6.89) | 11.52 (6.43)
  Change from Baseline Week 4: number analyzed (Participants) | 306 | 151
  Change from Baseline Week 4 | -6.51 (6.13) | -3.04 (5.04)
Statistical Analysis 1: Comparison: Elinzanetant (BAY3427080) vs Placebo - Elinzanetant (BAY3427080); Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM) — One-sided. A multiplicity adjustment strategy was defined using the hierarchical testing strategy, controlling the overall type I error rate at a one-sided alpha level of 0.025 for confirmatory statistical superiority testing; Diffrence in Least Squares (LS) means = -3.48, Standard Error of Mean 0.44

2. Primary Outcome: Mean Change in Frequency of Moderate to Severe HFs From Baseline to Week 12 (Assessed by HFDD)
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
hot flashes per day
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 11.41 (6.89) | 11.52 (6.43)
  Change from Baseline week 12: number analyzed (Participants) | 292 | 147
  Change from Baseline week 12 | -7.76 (6.17) | -4.20 (6.06)
Statistical Analysis 1: Comparison: Elinzanetant (BAY3427080) vs Placebo - Elinzanetant (BAY3427080); Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -3.38, Standard Error of Mean 0.43

3. Secondary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 4 (Assessed by HFDD).
Description: In the HFDD, the severity of HFs was categorized as: 1 = mild, 2 = moderate, and 3 = severe; therefore, a decrease in the HF severity score indicates an improvement.
  The mean daily severity during treatment was calculated for the available days as [(1 x number of mild HF) + (2 x number of moderate HF) + (3 x number of severe HF)] / (total number of mild, moderate and severe hot flashes on that day). When no HFs were reported for a particular day, the mean severity for that day was set to 0. The mean daily severity during baseline was calculated for the available days as [(2 x number of moderate HF) + (3 x number of severe HF)] / (total number of moderate to severe hot flashes on that day).
Time Frame: Baseline to Week 4
Population: FAS
Measure: Mean (Standard Deviation); unit: score*hot flashes/total of hot flashes
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
score*hot flashes/total of hot flashes
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 2.49 (0.24) | 2.49 (0.22)
  Change from Baseline week 4: number analyzed (Participants) | 306 | 151
  Change from Baseline week 4 | -0.73 (0.60) | -0.43 (0.43)

4. Secondary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 12 (Assessed by HFDD)
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: score*hot flashes/total of hot flashes
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
score*hot flashes/total of hot flashes
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 2.49 (0.24) | 2.49 (0.22)
  Change from Baseline week 12: number analyzed (Participants) | 292 | 147
  Change from Baseline week 12 | -0.98 (0.72) | -0.53 (0.60)

5. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 1 (Assessed by HFDD)
Description: as for outcome 1
Time Frame: Baseline to Week 1
Population: FAS
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
hot flashes per day
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 11.41 (6.89) | 11.52 (6.43)
  Change from baseline week 1: number analyzed (Participants) | 314 | 155
  Change from baseline week 1 | -4.04 (5.11) | -1.76 (3.83)

6. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline Over Time (Assessed by HFDD)
Description: as for outcome 1
Time Frame: Baseline to Week 50
Population: FAS
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
hot flashes per day
  Baseline: number analyzed (Participants) | 316 | 157
  Baseline | 11.41 (6.89) | 11.52 (6.43)
  Change from baseline to Week 1: number analyzed (Participants) | 314 | 155
  Change from baseline to Week 1 | -4.04 (5.11) | -1.76 (3.83)
  Change from baseline to Week 2: number analyzed (Participants) | 311 | 154
  Change from baseline to Week 2 | -5.55 (5.88) | -2.78 (4.31)
  Change from baseline to Week 3: number analyzed (Participants) | 311 | 154
  Change from baseline to Week 3 | -6.19 (5.94) | -2.96 (4.82)
  Change from baseline to Week 4: number analyzed (Participants) | 306 | 151
  Change from baseline to Week 4 | -6.51 (6.13) | -3.04 (5.04)
  Change from baseline to Week 5: number analyzed (Participants) | 302 | 149
  Change from baseline to Week 5 | -6.84 (5.92) | -3.35 (5.06)
  Change from baseline to Week 6: number analyzed (Participants) | 296 | 150
  Change from baseline to Week 6 | -7.04 (6.20) | -3.69 (5.37)
  Change from baseline to Week 7: number analyzed (Participants) | 297 | 148
  Change from baseline to Week 7 | -7.32 (6.05) | -3.96 (5.60)
  Change from baseline to Week 8: number analyzed (Participants) | 297 | 148
  Change from baseline to Week 8 | -7.45 (6.25) | -4.02 (5.53)
  Change from baseline to Week 9: number analyzed (Participants) | 294 | 149
  Change from baseline to Week 9 | -7.49 (6.29) | -4.00 (5.64)
  Change from baseline to Week 10: number analyzed (Participants) | 293 | 146
  Change from baseline to Week 10 | -7.48 (6.03) | -3.88 (5.82)
  Change from baseline to Week 11: number analyzed (Participants) | 293 | 149
  Change from baseline to Week 11 | -7.74 (6.16) | -4.08 (5.94)
  Change from baseline to Week 12: number analyzed (Participants) | 292 | 147
  Change from baseline to Week 12 | -7.76 (6.17) | -4.20 (6.06)
  Change from baseline to Week 25: number analyzed (Participants) | 272 | 135
  Change from baseline to Week 25 | -8.98 (6.12) | -9.60 (6.04)
  Change from baseline to Week 26: number analyzed (Participants) | 272 | 133
  Change from baseline to Week 26 | -8.93 (6.13) | -9.55 (6.14)
  Change from baseline to Week 35: number analyzed (Participants) | 265 | 134
  Change from baseline to Week 35 | -9.05 (6.16) | -9.30 (6.23)
  Change from baseline to Week 36: number analyzed (Participants) | 260 | 133
  Change from baseline to Week 36 | -8.94 (6.15) | -9.13 (6.25)
  Change from baseline to Week 49: number analyzed (Participants) | 255 | 127
  Change from baseline to Week 49 | -8.77 (5.89) | -9.02 (6.17)
  Change from baseline to Week 50: number analyzed (Participants) | 249 | 125
  Change from baseline to Week 50 | -8.72 (6.22) | -8.90 (6.01)

7. Secondary Outcome: Mean Change in Patient-reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total Score From Baseline to Week 12
Description: The PROMIS SD SF 8b includes 8 items assessing sleep disturbance over the past 7 days. Items assess sleep quality, sleep depth and restoration associated with sleep, perceived difficulties with getting to sleep or staying asleep and perceptions of the adequacy of and satisfaction with sleep. Participants respond to the items on a 5-point scale from "not at all", "never" or "very poor" to "very much", "always" or "very good". Four of the items are scored reversely. Individual item scores are aggregated to total raw scores which range from 8 to 40. Total raw scores are converted into T-scores for comparison with population norms, with a mean of 50 and standard deviation of 10. T-scores range from 28.9 to 76.5. For both raw and T-scores higher scores indicate greater severity of sleep disturbance. According to available score cut points from PROMIS developers, T-scores can be interpreted as indicating mild (55-59), moderate (60-69), or severe (>70) sleep disturbance.
Time Frame: Baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
T-Score
  Baseline: number analyzed (Participants) | 313 | 155
  Baseline | 60.60 (6.33) | 60.74 (6.80)
  Change from Baseline week 12: number analyzed (Participants) | 289 | 146
  Change from Baseline week 12 | -10.55 (8.20) | -4.06 (7.35)
Statistical Analysis 1: Comparison: Elinzanetant (BAY3427080) vs Placebo - Elinzanetant (BAY3427080); Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in Least Squares Means = -6.12, Standard Error of Mean 0.70

8. Secondary Outcome: Mean Change in Menopause Specific Quality of Life Scale (MENQOL) Total Score From Baseline to Week 12
Description: The MENQOL questionnaire is comprised of 29 items assessing the presence of menopausal symptoms and the impact of menopause on health-related quality of life over the past week. The items assess four domains of symptoms and functioning: VMS, psychosocial functioning, physical functioning, and sexual functioning. For each item, the participant indicates if they have experienced the symptom (yes/no). If participants select yes, participants rate how bothered they were by the symptom using a six-point verbal descriptor scale, with response options ranging from 0 'not at all bothered' to 6 'extremely bothered'. Based on the individual responses, item scores, domain scores, and a total MENQOL score are calculated. Each score ranges from 1-8, higher scores indicate greater bother. For a MENQOL total score, the aggregated mean of the mean domain scores is calculated.
Time Frame: Baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant (BAY3427080) | Placebo - Elinzanetant (BAY3427080)
Number analyzed (Participants) | 316 | 158
Scores on a scale
  Baseline: number analyzed (Participants) | 311 | 155
  Baseline | 4.82 (1.17) | 4.77 (1.25)
  Change from Baseline week 12: number analyzed (Participants) | 285 | 143
  Change from Baseline week 12 | -1.30 (1.11) | -0.53 (1.15)
Statistical Analysis 1: Comparison: Elinzanetant (BAY3427080) vs Placebo - Elinzanetant (BAY3427080); Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in Last Squares Means = -0.68, Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: From signing the ICF through study complition, approximately 14 months
Groups:
- Elinzanetant 120mg Week 1-12: Participants who received elinzanetant 120 mg during Weeks 1-12. Only AEs that were reported during Weeks 1-12 are included in the safety tables.
- Placebo Week 1-12: Participants who received placebo during Weeks 1-12. Only AEs that were reported during Weeks 1-12 are included in the safety tables.
- Elinzanetant 120mg Week 13-26: Participants who received elinzanetant 120 mg during Week 1-12 and continued elinzanetant 120 mg after Week 12. Only AEs that were reported during Weeks 13-26 are included.
- Placebo - Elinzanetant 120mg Week 13-26: Participants who received placebo during Weeks 1-12 and switched to elinzanetant 120 mg after Week 12. Only AEs that were reported during Weeks 13-26 are included.
- Elinzanetant 120mg Week 1-26: Participants who received elinzanetant 120 mg during Weeks 1-26 (including those who switched from placebo to elinzanetant 120 mg at Week 13). AEs that were reported during placebo period (Weeks 1-12) are excluded.
- Elinzanetant 120mg Week 27-52: Participants who received elinzanetant 120 mg during Weeks 27-52. Only AEs that were reported during Weeks 27-52 are included.
- Elinzanetant 120mg Week 1-52: Participants who received elinzanetant 120 mg at any time during the study (including those who switched from placebo to elinzanetant 120 mg at Week 13). AEs that were reported during placebo period (Weeks 1-12) are excluded.
Arm/Group | Elinzanetant 120mg Week 1-12 | Placebo Week 1-12 | Elinzanetant 120mg Week 13-26 | Placebo - Elinzanetant 120mg Week 13-26 | Elinzanetant 120mg Week 1-26 | Elinzanetant 120mg Week 27-52 | Elinzanetant 120mg Week 1-52
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/158 | 0/294 | 0/150 | 0/465 | 0/409 | 0/465
Serious Adverse Events (participants affected / at risk) | 8/315 | 1/158 | 8/294 | 4/150 | 18/465 | 18/409 | 33/465
Other Adverse Events (participants affected / at risk) | 145/315 | 61/158 | 72/294 | 38/150 | 211/465 | 73/409 | 241/465
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120mg Week 1-12 (N=315) | Placebo Week 1-12 (N=158) | Elinzanetant 120mg Week 13-26 (N=294) | Placebo - Elinzanetant 120mg Week 13-26 (N=150) | Elinzanetant 120mg Week 1-26 (N=465) | Elinzanetant 120mg Week 27-52 (N=409) | Elinzanetant 120mg Week 1-52 (N=465)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anisomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometrial hyperplasia with cellular atypia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ligament operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120mg Week 1-12 (N=315) | Placebo Week 1-12 (N=158) | Elinzanetant 120mg Week 13-26 (N=294) | Placebo - Elinzanetant 120mg Week 13-26 (N=150) | Elinzanetant 120mg Week 1-26 (N=465) | Elinzanetant 120mg Week 27-52 (N=409) | Elinzanetant 120mg Week 1-52 (N=465)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 3 (3) | 6 (6) | 4 (4) | 25 (29) | 7 (7) | 32 (36)
Nausea (Gastrointestinal disorders) | 19 (20) | 10 (12) | 6 (6) | 5 (7) | 28 (33) | 3 (3) | 29 (36)
Asthenia (General disorders) | 13 (14) | 2 (2) | 7 (7) | 3 (3) | 22 (24) | 5 (5) | 26 (30)
Fatigue (General disorders) | 30 (37) | 8 (10) | 7 (7) | 5 (7) | 41 (51) | 3 (3) | 43 (57)
COVID-19 (Infections and infestations) | 4 (4) | 4 (4) | 9 (9) | 4 (6) | 17 (19) | 13 (13) | 32 (34)
Nasopharyngitis (Infections and infestations) | 12 (13) | 5 (5) | 9 (10) | 8 (8) | 28 (31) | 9 (10) | 37 (41)
Depression rating scale score increased (Investigations) | 21 (21) | 13 (14) | 1 (1) | 0 (0) | 22 (22) | 2 (2) | 26 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 10 (10) | 19 (21) | 6 (6) | 42 (49) | 15 (15) | 52 (65)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 7 (10) | 5 (5) | 2 (2) | 16 (17) | 14 (14) | 29 (31)
Headache (Nervous system disorders) | 30 (42) | 20 (24) | 13 (17) | 7 (8) | 48 (67) | 11 (16) | 56 (85)
Somnolence (Nervous system disorders) | 34 (37) | 6 (6) | 4 (4) | 5 (5) | 42 (46) | 1 (1) | 42 (47)
Depression (Psychiatric disorders) | 14 (14) | 1 (1) | 7 (7) | 2 (2) | 23 (23) | 5 (5) | 28 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05587296/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT05587296/SAP_001.pdf